CLINICAL TRIAL: NCT06216795
Title: Measurement of Kidney Volume Using Computed Tomography in Kidney Transplant Donors and Recipients
Brief Title: Kidney Volume in Live Donors Kidney Transplant Donors and Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUH-Kidney Volumetry_KT_v1.3
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Kidney Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- kidney transplant group

SUMMARY:
The investigators aim to investigate the association between renal volume measured through pre-donation CT auto-segmentation and postoperative renal function of both donors and recipients. After establishing the statistical significance of the association, the investigators intend to create and validate predictive models for renal function at surgery, 1 year, and 3 years postoperatively, incorporating various factors known to contribute to renal function deterioration.

ELIGIBILITY:
Inclusion Criteria:

* live donor kidney transplant

Exclusion Criteria:

* donors without preoperative enhanced CT image

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: live kidney donors and paired their recipients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction models for the residual renal function of donors and the graft kidney function of recipient after live donor kidney transplantation | 1 and 3 years after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jo EA, Lee J, Moon S, Kim JS, Han A, Ha J, Kim YC, Min S. The role of artificial intelligence measured preoperative kidney volume in predicting kidney function loss in elderly kidney donors: a multicenter cohort study. Int J Surg. 2024 Nov 1;110(11):7169-7176. doi: 10.1097/JS9.0000000000002030. PMID 39116451